CLINICAL TRIAL: NCT03421119
Title: A Phase III, Randomized, Parallel, Double-blind, and Non-inferiority Clinical Trial to Compare Efficacy and Safety of CinnaGen-liraglutide to Innovator Liraglutide Product (Victoza®) in Patients With Type II Diabetes (T2D)
Brief Title: Comparing Efficacy and Safety of CinnaGen-liraglutide Versus Victoza® in Patients With Type II Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIR.CIN.MK95
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; liraglutide; efficacy; safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CinnaGen-liraglutide (Experimental): CinnaGen-liraglutide (Liraglutide 6 MG/ML Pen Injector by CinnaGen Company) will be administered 1.8 mg/day subcutaneously. Doses of CinnaGen-liraglutide will be up-titrated from 0.6 mg/day in the first week to 1.2 mg/day in the second, third and fourth weeks, up to 1.8 mg/day from the start of the fifth week to the end of 26th week. Patients in this group will continue to receive metformin along with a Sulfonylurea/non-sulfonylurea insulin secretagogues with maximum tolerable dose.
  Interventions: Drug: Liraglutide 6 MG/ML Pen Injector; Drug: Metformin; Drug: Sulfonylurea/non-sulfonylurea insulin secretagogues
- Victoza® (Active Comparator): Victoza® (Liraglutide 6 MG/ML Pen Injector by Novo Nordisk Company) will be administered 1.8 mg/day subcutaneously. Doses of Victoza® will be up-titrated from 0.6 mg/day in the first week to 1.2 mg/day in the second, third and fourth weeks, up to 1.8 mg/day from the start of the fifth week to the end of 26th week. Patients in this group will continue to receive metformin along with a Sulfonylurea/non-sulfonylurea insulin secretagogues with maximum tolerable dose.
  Interventions: Drug: Liraglutide 6 MG/ML Pen Injector; Drug: Metformin; Drug: Sulfonylurea/non-sulfonylurea insulin secretagogues

INTERVENTIONS:
Drug: Liraglutide 6 MG/ML Pen Injector — Patients in each arm will receive either CinnaGen-liraglutide or Victoza®. Both products will be provided as pen-injector.
  Other Names: CinnaGen-liraglutide, Victoza
Drug: Metformin — Patients who were receiving metformin with maximum tolerable dose prior to study will continue to receive it during the study.
  Other Names: Metformin Hydrochloride
Drug: Sulfonylurea/non-sulfonylurea insulin secretagogues — Patients who were receiving Sulfonylurea/non-sulfonylurea insulin secretagogues with maximum tolerable dose prior to study will continue to receive it during the study.
  Other Names: Sulfonylurea or non-sulfonylurea insulin secretagogues

SUMMARY:
The purpose of this study is to compare the efficacy and safety of liraglutide produced by CinnaGen company and Novo Nordisk liraglutide (Victoza®) in subjects with type II diabetes. Patients with Type II diabetes treated with two oral glucose-lowering agents for ≥ 3 months, aged between 30 to 65 years, HbA1c equal or greater than 7.5 and lower than 10, and BMI between 25 to 45 were included in this study.

This study is a phase III, randomized, two-armed, parallel, double-blind, active-controlled, and non-inferiority clinical trial. Patients who enter the trial will be randomly allocated (1:1 ratio) to receive subcutaneous 1.8 mg daily injections of either Victoza® or CinnaGen-liraglutide. Doses of liraglutide will be up-titrated from 0.6 mg/day in the first week to 1.2 mg/day in the second, third and fourth weeks up to 1.8 mg/day from the beginning of the fifth week. Patients continue to receive 1.8 mg/day liraglutide until the end 26th week.

The primary objective of this study is to assess non-inferiority of CinnaGen-liraglutide to reference liraglutide in terms of efficacy in patients with T2D. The secondary objectives of this study are to further compare the efficacy of CinnaGen-liraglutide to reference liraglutide and to assess the safety of CinnaGen-liraglutide to reference liraglutide.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and safety of liraglutide produced by CinnaGen company with Novo Nordisk liraglutide (Victoza®) in subjects with type II diabetes. Patients with Type II diabetes treated with two oral glucose-lowering agents for ≥ 3 months, aged between 30 to 65 years, HbA1c equal or greater than 7.5 and lower than 10, and BMI between 25 to 45 will be included in this study. This study is a phase III, randomized, two-armed, parallel, double-blind, active-controlled, and non-inferiority clinical trial. Patients who enter the trial will be randomly allocated (1:1 ratio) to receive subcutaneous 1.8 mg daily injections of either Victoza® or CinnaGen-liraglutide. Doses of liraglutide will be up-titrated from 0.6 mg/day in the first week to 1.2 mg/day in the second, third and fourth weeks up to 1.8 mg/day from the beginning of the fifth week. Patients continue to receive 1.8 mg/day liraglutide until the end of 26th week.

Physical examinations and vital signs will be evaluated for patients at baseline, and at weeks 4, 8, 12 and 26 visits. Laboratory parameters will be assessed at baseline, week 12 and 26. The incidence of adverse events will be evaluated based on patients' reports, vital signs, physical examinations, and laboratory tests.

Before initiation, the trial will be reviewed by food and drug administration of Iran. The protocol, electronic case report form (eCRF), information for patients and informed consent form will be submitted to the ethics committees responsible for review and approval purposes, according to national regulatory guidelines.

In this study, no patient will be recruited without informed consent. All the informed consent forms which will be signed by the patients will have two copies so that patients can receive a copy of it.

Determination of sample size:

Group sample sizes of 120 and 120 achieve 80% power to detect non-inferiority using a one-sided, two-sample t-test with a non-inferiority margin of -0.4. The true difference between the means is assumed to be zero. The significance level (alpha) of the test is 0.025. The data are drawn from populations with standard deviations of 1.1 and considering a drop-out rate of 20% total sample size required is 300 patients.

Data Quality Assurance:

CinnaGen Company conducts clinical trials according to procedures that incorporate the ethical principles of GCP. Accurate and reliable data collection is assured by verification and cross-check of the eCRFs against the patient's records by clinical monitors, and the maintenance of a drug-dispensing log by the center.

CRO coordinators and sponsor attend the SIV (Site Initiation Visit) meetings. Protocol and GCP principles will be reviewed by coordinating investigator of each site, and also the needed information for completing eCRF forms will be explained.

Monitoring by CRO is performed in 30% and 70% of study progress and at the end of the study. In the monitoring sessions some sponsor personnel audit the process. During the monitoring process, CRO coordinator checks all eCRFs and confirms them to the source documents, and for required cases, the query form will be filled out.

The temperature of the refrigerator containing the medicines is checked and recorded by data logger which will be monitored regularly by the auditor.

CRO coordinator will verify drug accountability data and information about the proper time for patients' injections, and sponsor staff rechecks it.

After monitoring, problems are reported by monitor and auditor to the trial centers.

Blinding:

In order to prevent the influence of knowing intervention group on study results, the patients and those who assess the study outcomes will remain unaware of allocation to test- or reference-liraglutide.

For this purpose, patients and caregivers will be masked to allocated treatment by making reference and test products indiscernible by appearance. Medicines will be provided in a similar dosage form labeled with a unique code.

It should be noted that CRO personnel who enter data into eCRF and database and also the sponsoring personnel who monitor data entry are blinded. The study is double-blind and situations that might warrant breaking the code are defined in the protocol and include serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes treated with maximum tolerable dose of two oral glucose-lowering agents (OGLAs; Metformin along with a Sulfonylurea/non-sulfonylurea insulin secretagogues) for ≥ 3 months
* 30-65 years of age
* 7.5 ≤ HbA1c < 10
* Body mass index (BMI) of 25-45 kg / m2

Exclusion Criteria:

* Lack of consent for being in the trial and not complying with 26-weeks follow-up period;
* Hypersensitivity to liraglutide or any component of the formulation (excipients include Disodium phosphate dehydrate, Propylene glycol, Phenol, Water for injection)
* Insulin treatment during the previous 3 months (except short-term treatment for intercurrent illness)
* Impaired liver function (alanine aminotransferase concentrations ≥ 2·5 times upper normal range).
* Impaired renal function (eGFR < 60 mL/min/1.73 m2),
* Uncontrolled hypertension (≥ 160/100 mmHg),
* Malignancy
* Used any drugs apart from OGLAs likely to affect glucose concentrations, including androgens, hyperglycemia-associated agents, hypoglycemia-associated agents, MAO inhibitors, quinolone antibiotics, salicylates (Anti-inflammatory dose).
* Treatment with dipeptidyl peptidase 4 inhibitors (DPP4 inhibitors)
* Treatment with systemic corticosteroids
* History or family history of Medullary Thyroid Carcinoma (MTC)
* Multiple endocrine neoplasia syndrome type 2 (MEN2)
* History of pancreatic cancer and pancreatitis
* History of recent MI, uncontrolled CHF, and unstable Angina
* History or known case of severe non-proliferative diabetic retinopathy or proliferative diabetic retinopathy
* Pregnancy
* Previous exposure to exenatide or liraglutide

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 26 weeks
  The primary outcome of this study is to assess changes in HbA1c in both treatment arms

SECONDARY OUTCOMES:
HbA1c < 7.0% | 26 weeks
  Percentages of subjects achieving HbA1c < 7.0% is measured in both treatment arms
HbA1c ≤ 6.5% | 26 weeks
  Percentages of subjects achieving HbA1c ≤ 6.5% is measured in both treatment arms
Body weight | 26 weeks
  Changes in body weight is measured in both treatment arms
Fasting blood sugar | 26 weeks
  Changes in FBS is measured in both treatment arms
Postprandial glucose | 26 weeks
  Changes in mean PPG is measured in both treatment arms
Systolic blood pressure | 26 weeks
  Changes in SBP (mmHg) is measured in both treatment arms
Diastolic blood pressure | 26 weeks
  Changes in DBP (mmHg) is measured in both treatment arms
Lipid profiles | 26 weeks
  Changes in Lipid profiles is measured in both treatment arms
Pulse Rate | 26 weeks
  Changes in PR is measured in both treatment arms
estimated Glomerular Filtration Rate | 26 weeks
  Changes in eGFR is measured in both treatment arms
Liver enzymes | 26 weeks
  Changes in AST and ALT is measured in both treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ebrahim Khamseh, Professor, Principal Investigator — Endocrine Research Center, Institute of Endocrinology and Metabolism, Iran University of Medical Sciences, Tehran, Iran.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nauck M, Frid A, Hermansen K, Shah NS, Tankova T, Mitha IH, Zdravkovic M, During M, Matthews DR; LEAD-2 Study Group. Efficacy and safety comparison of liraglutide, glimepiride, and placebo, all in combination with metformin, in type 2 diabetes: the LEAD (liraglutide effect and action in diabetes)-2 study. Diabetes Care. 2009 Jan;32(1):84-90. doi: 10.2337/dc08-1355. Epub 2008 Oct 17. PMID 18931095
- [Background] Marre M, Shaw J, Brandle M, Bebakar WM, Kamaruddin NA, Strand J, Zdravkovic M, Le Thi TD, Colagiuri S; LEAD-1 SU study group. Liraglutide, a once-daily human GLP-1 analogue, added to a sulphonylurea over 26 weeks produces greater improvements in glycaemic and weight control compared with adding rosiglitazone or placebo in subjects with Type 2 diabetes (LEAD-1 SU). Diabet Med. 2009 Mar;26(3):268-78. doi: 10.1111/j.1464-5491.2009.02666.x. PMID 19317822
- [Background] Zinman B, Gerich J, Buse JB, Lewin A, Schwartz S, Raskin P, Hale PM, Zdravkovic M, Blonde L; LEAD-4 Study Investigators. Efficacy and safety of the human glucagon-like peptide-1 analog liraglutide in combination with metformin and thiazolidinedione in patients with type 2 diabetes (LEAD-4 Met+TZD). Diabetes Care. 2009 Jul;32(7):1224-30. doi: 10.2337/dc08-2124. Epub 2009 Mar 16. PMID 19289857
- [Background] Russell-Jones D, Vaag A, Schmitz O, Sethi BK, Lalic N, Antic S, Zdravkovic M, Ravn GM, Simo R; Liraglutide Effect and Action in Diabetes 5 (LEAD-5) met+SU Study Group. Liraglutide vs insulin glargine and placebo in combination with metformin and sulfonylurea therapy in type 2 diabetes mellitus (LEAD-5 met+SU): a randomised controlled trial. Diabetologia. 2009 Oct;52(10):2046-55. doi: 10.1007/s00125-009-1472-y. Epub 2009 Aug 14. PMID 19688338
- [Background] Buse JB, Rosenstock J, Sesti G, Schmidt WE, Montanya E, Brett JH, Zychma M, Blonde L; LEAD-6 Study Group. Liraglutide once a day versus exenatide twice a day for type 2 diabetes: a 26-week randomised, parallel-group, multinational, open-label trial (LEAD-6). Lancet. 2009 Jul 4;374(9683):39-47. doi: 10.1016/S0140-6736(09)60659-0. Epub 2009 Jun 8. PMID 19515413
- [Derived] Esteghamati A, Zamanzadeh M, Malek M, Khaledi M, Monavari A, Najafi L, Banazadeh Z, Malboosbaf R, Aghili R, Mahdikhah S, Ganjizadeh-Zavereh H, Kafi H, Hosseinpanah F, Khamseh ME. Efficacy and Safety of a Biosimilar Liraglutide (Melitide(R)) Versus the Reference Liraglutide (Victoza(R)) in People with Type 2 Diabetes Mellitus: A Randomized, Double-Blind, Noninferiority Clinical Trial. Diabetes Ther. 2023 Nov;14(11):1889-1902. doi: 10.1007/s13300-023-01462-w. Epub 2023 Sep 14. PMID 37707701